CLINICAL TRIAL: NCT00149760
Title: Cognitive Affective Behavior Therapy for Somatization
Brief Title: Effectiveness of Cognitive-Affective Behavior Therapy for the Treatment of Somatization Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21MH066831 (NIH); R21MH066831 (NIH); DAHBR 96-BHC
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Somatization Disorder
Keywords: Cognitive Behavior Therapy; Treatment Outcome; Health Care Utilization; Somatization Disorder; Somatoform Disorder
MeSH Terms: conditions — Somatoform Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmented Standard Medical Care (Active Comparator): Participants will receive standard medical care augmented by a psychiatric consultation letter sent to the participants' primary care physician.
  Interventions: Behavioral: Augmented Standard Medical Care
- Cognitive-Affective Behavior Therapy (Experimental): Participants will receive individually administered cognitive-affective behavior therapy as well as augmented standard medical care.
  Interventions: Behavioral: Cognitive-Affective Behavior Therapy

INTERVENTIONS:
Behavioral: Augmented Standard Medical Care — Participants' physicians will receive a letter making specific treatment recommendations for primary care treatment.
  Other Names: Psychiatric consultation letter sent to primary physician
  Arms: Augmented Standard Medical Care
Behavioral: Cognitive-Affective Behavior Therapy — Individually-administered cognitive-behavioral therapy with an emotional focus in addition to augmented standard medical care
  Other Names: Emotionally-Focused Cognitive-Behavioral Therapy
  Arms: Cognitive-Affective Behavior Therapy

SUMMARY:
This study will examine the long-term effect of cognitive-affective behavior therapy on the physical symptoms, functioning, and health care utilization of people with somatization disorder.

DETAILED DESCRIPTION:
Somatization disorder is a syndrome characterized by the presence of multiple medically unexplained physical symptoms. It often results in substantial functional impairment and the need for extensive medical treatment. Neither pharmacological nor psychosocial treatments for the disease have demonstrated clinical success. People with somatization disorder may benefit from a treatment that integrates emotion-centered strategies into cognitive behavioral therapy. The long-term effectiveness of this treatment has not been established, however. This study will examine the long-term effect of cognitive-affective behavior therapy on the physical symptoms, functioning, and health care utilization of people with somatization disorder.

Participants in this open-label study will be randomly assigned to receive either cognitive-affective behavior therapy (CABT) or standard medical care that is augmented by a psychiatric consultation. Treatment will last 4 months. Assessments of somatic symptomatology, functional impairment, and health care costs will occur at screening, baseline (1 to 2 weeks after screening), and 4, 10, and 16 months after baseline. The visits at 10 and 16 months post-baseline will assess specifically the long-term efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for somatization disorder
* Available for follow-up over the ensuing 18 months
* English-speaking

Exclusion Criteria:

* Meets DSM-IV criteria for a psychotic disorder, organic brain syndrome, or psychoactive substance dependence (Other psychiatric comorbidity is not exclusionary)
* Active suicidal ideation
* Unstable major medical condition
* Plans to engage in additional psychotherapy during the first 6 months after enrollment
* Current use of any medication that has not been stabilized for the previous 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale for Somatization Disorder | Measured at baseline and Months 4, 10, and 16

SECONDARY OUTCOMES:
Physical functioning | Measured at baseline and Months 4, 10, and 16
Health care utilization | Measured between Months 4 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A. Allen, PhD, Principal Investigator — Department of Psychiatry, Robert Wood Johnson Medical School
Locations (1):
- Department of Psychiatry, Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

REFERENCES:
- [Background] Allen LA, Woolfolk RL, Lehrer PM, Gara MA, Escobar JI. Cognitive behavior therapy for somatization disorder: a preliminary investigation. J Behav Ther Exp Psychiatry. 2001 Jun;32(2):53-62. doi: 10.1016/s0005-7916(01)00020-9. PMID 11764061
- [Background] Allen LA, Escobar JI, Lehrer PM, Gara MA, Woolfolk RL. Psychosocial treatments for multiple unexplained physical symptoms: a review of the literature. Psychosom Med. 2002 Nov-Dec;64(6):939-50. doi: 10.1097/01.psy.0000024231.11538.8f. PMID 12461199
- [Background] Allen, Lesley A. Short-term therapy for somatization disorder: A cognitive behavioral approach. Journal of Cognitive Psychotherapy. Vol 14(4) Win 2000, 373-380.
- [Background] Allen LA, Woolfolk RL, Escobar JI, Gara MA, Hamer RM. Cognitive-behavioral therapy for somatization disorder: a randomized controlled trial. Arch Intern Med. 2006 Jul 24;166(14):1512-8. doi: 10.1001/archinte.166.14.1512. PMID 16864762